CLINICAL TRIAL: NCT03372304
Title: Catheter-based Peripheral Regional Anesthesia After Orthopedic Surgery to the Foot or Ankle: Comparison of Low Dose, Automated Periodic Infusions With Conventional High Dose, Continuous Infusion, and Patient-initiated Infusions Only
Brief Title: Catheter-based Peripheral Regional Anesthesia After Orthopedic Surgery to the Foot or Ankle
Acronym: API-FOOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Principal Investigator, Claus Behrend Christiansen, Medical doctor, Nordsjaellands Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-17021730
Record Dates: First submitted 2017-12-10; First posted 2017-12-13 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Pain
Keywords: Peripheral regional anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: 3 arms (API, CI and PCA only)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All patients and outcome assessors will be blinded to the delivery administrations. Investigators will not be present while programming of the infusion pump is taking place. The display of the infusion pump will be concealed at all times after initiation. Furthermore, throughout the trial, the infusion pump will be concealed from the patient through a non-transparent bag. Trial interventions will not be visible in electronic patient charts. The infusion pump is making a discrete noise when administering medications. To make sure that the PCA group and the continuous infusion group is blinded to interventions, a sham administration is activated every 8th hour. This sham administration will be 0.1 mL of ropivacaine 0.2%. Such a small dose of LA will not have any anesthetic effect nor pose a risk for the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- API+PCA (Experimental): Infusion of ropivacaine 0.2 %, 10 mL, every 8th hour. Patient-initiated bolus of ropivacaine 0.2 %, 10 mL. Lock-out time: 4 hours.
  Interventions: Drug: Ropivacaine 0.2%
- CI+PCA (Active Comparator): Continuous infusion of ropivacaine 0.2 %, 6 mL/hour. Patient-initiated bolus of ropivacaine 0.2 %, 10 mL. Lock-out time: 4 hours.
  Interventions: Drug: Ropivacaine 0.2%
- PCA only (Active Comparator): Patient-initiated bolus of ropivacaine 0.2 %, 10 mL. Lock-out time: 4 hours.
  Interventions: Drug: Ropivacaine 0.2%

INTERVENTIONS:
Drug: Ropivacaine 0.2% — Perineural infusion of Ropivacaine 0.2% using a peripheral nerve block catheter and a portable infusion pump.
  Other Names: Naropin 0.2%

SUMMARY:
BACKGROUND

Orthopedic surgery can be severely painful, and peripheral regional anesthesia is highly recommended as part of the perioperative pain treatment. Whether catheter-based techniques are better than single injection techniques are debatable. Furthermore, in catheter-based techniques, whether a low-dose automated, periodic infusion can produce similar analgesic effectiveness compared to a conventional, high dose, continuous infusion has never been explored.

AIM

Comparison of the analgesic effectiveness of a low-dose automated, periodic infusion, a conventional continuous infusion and patient-controlled boluses only in catheter-based nerve blocks for patients undergoing orthopedic surgery to the foot or ankle.

DETAILED DESCRIPTION:
BACKGROUND

Orthopedic surgery has been reported to be moderate to severely painful in approximately 50 % of patients.

Peripheral regional anesthesia (PRA) using single injection nerve blocks is highly recommended as part of a multimodal, perioperative, analgesic treatment. Patients who are expected to have postoperative, severe pain exceeding the duration of a single injection nerve block may benefit from a catheter-based nerve block (CBNB) using either a continuous infusion (CI) or intermittent infusions of local anesthetics (LA). Intermittent boluses can be either patient-controlled or prescribed in combination with a continuous infusion or as prespecified intermittent boluses. Whether a CBNB treatment is superior to a single injection nerve block after orthopedic surgery remains unanswered.

There are several challenges when using a CBNB treatment: The dosing or delivery method may be either insufficient and thus not pain relieving or too powerful resulting in dense motor block and limb anesthesia which may compromise safety and rehabilitation. The peripheral nerve block catheter may also displace and therefore deposit LA too far from the targeted nerve(s) to produce an effective nerve block.

Previous studies suggest that an automated periodic infusion (API) regimen is superior to CI. It seems that an API produces better pain control, a lower analgesic consumption over time and less motor inhibition. This is well-described for epidural catheters for laboring women, but evidence is also apparent in PRA. Adding a PCA bolus option to a catheter-based nerve block treatment may even out the difference in pain scores between API and CI. However, it seems that API groups require less LA via PCA function. Reducing LA consumption is of great importance for ambulatory patients whose LA reservoir is limited, but also for all other orthopedic patients whose motor block should be minimized in order to optimize rehabilitation.

OBJECTIVES

To investigate whether a low-dose API with patient-controlled bolus option can produce a similar analgesic effect compared to a conventional, high dose, CI with patient-controlled bolus option in catheter-based peripheral nerve blocks for patients undergoing orthopedic surgery to the foot or ankle. Analgesic effectiveness will be compared with a group only given the patient-controlled bolus option.

HYPOTHESIS

Low dose API with supplemental patient-controlled bolus option will provide pain-relieving therapy not inferior to a conventional CI with supplemental patient-controlled bolus option. The intervention group receiving patient-controlled boluses only will experience more pain breakthrough.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists Classification I-III
2. Normal cognitive function in order to sign written, informed consent and to understand trial protocol
3. Agreement to the trial protocol, including the randomized manner

Exclusion Criteria:

1. Allergy to LA
2. Infection in or near insertion site of the peripheral nerve catheter
3. Anatomical abnormalities preventing successful peripheral nerve catheter insertion
4. Habitual use of opioids
5. Pregnancy or breastfeeding (disproved by a negative pregnancy test before trial inclusion)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Postoperative pain, 1-72 hours postoperatively | 1-72 hours
  Postoperative pain using the visual analogue pain scale (VAS, 0-100 milimetres). Measurements will be patient-reported.

SECONDARY OUTCOMES:
Opioid consumption, 1-72 hours postoperatively | 1-72 hours
  Tablets consumed during the period of investigation
Volume of patient-initiated boluses, 1-72 hours postoperatively | 1-72 hours
  Volume of ropivacaine 0.2 % (mL) used for patient-initiated boluses, 1-72 hours postoperatively

OTHER OUTCOMES:
Opioid related side effects | 1-72 hours
  Patient reported symptoms: dizziness, nausea, itching, constipation
Pain at bolus request | 1-72 hours
  Pain (VAS, 0-100 milimetres) at the time of patient-initiated bolus
Motor nerve block | 1-72 hours
  Degree of motor nerve block, defined by paresis or paralysis in the ankle dorsi- and plantarflexion movement.
Sensory nerve block | 1-72 hours
  Insensitivity towards cold in the lateral aspects of the lower leg and beneath the foot. This will be recorded by the patient using a cold glass vial stored in a refrigerator until its use.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Henrik Wiborg Lange, DMSci, Study Director — Department of Anesthesiology, Nordsjaellands Hospital & University of Copenhagen
Locations (1):
- Department of Anesthesiology, Nordsjællands Hospital Hillerød, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Undecided